CLINICAL TRIAL: NCT00833742
Title: Emotion-focused Diagnosis and Treatment of Somatization in the ED
Brief Title: Intensive Short-term Dynamic Psychotherapy (ISTDP) in the Emergency Department
Acronym: ISTDPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA01
Record Dates: First submitted 2008-02-12; First posted 2009-02-02 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2009-01

CONDITIONS: Somatic Complaints of Multiple Types
Keywords: somatization; psychosomatic; short-term; dynamic; psychotherapy
MeSH Terms: interventions — Psychotherapy, Brief

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ISTDP therapy was provided
  Interventions: Behavioral: Intensive Short-term Dynamic Psychotherapy
- 2 (No Intervention): People referred but never seen

INTERVENTIONS:
Behavioral: Intensive Short-term Dynamic Psychotherapy — A brief psychotherapy format
  Other Names: Short-term Psychotherapy
  Arms: 1

SUMMARY:
Objective: Somatization of emotions accounts for excess Emergency department (ED) visits. Intensive Short-term Dynamic Psychotherapy (ISTDP) has methods to diagnose and manage somatization. We examined the feasibility, acceptability and effectiveness of ISTDP diagnostic and treatment methods used for patients with repeated ED presentations for medically unexplained physical symptoms (MUS)

DETAILED DESCRIPTION:
Herein we report the methods and outcomes of rapidly-accessed, emotion-focused diagnostic and treatment services for patients presenting to the ED with medically unexplained symptoms (MUS). Patients who were assessed and referred by ED physicians will serve as a non-randomized condition controlling for some relevant variables. Our a priori hypotheses were that assessed and treated patients would have a reduction in ED visits and self reported symptoms after this intervention and that controls would have a smaller reduction in ED visits if any.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained symptoms

Exclusion Criteria:

* Psychosis, substance abuse, suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2002-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Emergency department visits pre and post | 1 year

SECONDARY OUTCOMES:
Brief Symptom Inventory | pre and post
Patient Satisfaction | post

CONTACTS AND LOCATIONS:
Overall Officials: Allan A Abbass, MD FRCPC, Principal Investigator — Capital Health, Canada
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Abbass A. Somatization: Diagnosing it sooner through emotion-focused interviewing. J Fam Pract. 2005 Mar;54(3):231-9, 243. No abstract available. PMID 15755376